CLINICAL TRIAL: NCT06774690
Title: Intra Artherial Therapies in Treatment of Primary Liver Diseases: an Observational Study
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: IAT for liver cancer
Record Dates: First submitted 2025-01-09; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-10

CONDITIONS: HCC - Hepatocellular Carcinoma; Cholangiocarcinoma Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 9 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to learn what are the best conditions that will give a positive outcome to men and women that receive a intra arterial therapy (IAT) for primary liver cancer.

Intra arterial therapies are radiologic procedures that block liver cancer blood supply.

The researchers will collect the data of participants located in the Radiology department in "IRCCS Azienda Ospedaliera Universitaria" Hospital in Bologna and will study clinic and radiological traits to understand which is the best case scenario for a optimal treatment response.

DETAILED DESCRIPTION:
This study is non profit, observational, retrospective, prospective and single institution.

The researchers will do a retrospective and prospective data collection and analyze the results. They will examine the radiological images (CT scan and RM) to assess the type and size of the cancer, track how the disease responds to treatments, identify possible complications.

There are no drugs involved and all the intra arterial therapies are performed within the routine clinical-care path.

* For the retrospective phase the researchers will analyze radiological image of the participants that received a intra arterial therapy from the 1st of January 2009. It's expected to enroll around 2000 participants.
* For the prospective phase the researchers will enroll for 5 years eligible participants that will receive a intra arterial therapy. Participants will go through a follow up every three months for the duration of the whole study. It is expected to enroll around 1300 participants.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Hepatocellular carcinoma (HCC) or intrahepatic cholangiocarcinoma (iCCA) and clinical indication to receive or have already received one of the following treatments:

  * Trans-arterial embolization (TAE),
  * Transarterial chemoembolization (TACE),
  * Transarterial radioembolization (TARE)
  * Drug-eluting beads chemoembolization (DEB-TACE)
* Age over 18
* To give informed consent

Exclusion Criteria:

* shunt of gastro intestinal arteries that cannot be embolized
* metastasis spread outside of the liver
* liver failure

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The participants will be selected from patients that are followed at Radiology Department of IRCCS Azienda Ospedaliero-Universitaria hospital in the city of Bologna.
Sampling Method: Non-Probability Sample
Enrollment: 3300 (Estimated)
Dates: Start 2021-04-21 (Actual); Primary Completion 2030-03 (Estimated); Study Completion 2030-04 (Estimated)

PRIMARY OUTCOMES:
Type and size of the injury | From enrollment to the end of treatment at 9 years
  Type and size of the injury
Radiological response to therapy | From enrollment to the end of treatment at 9 years
  Radiological response to therapy
Post treatment complications | From enrollment to the end of treatment at 9 years
  Post treatment complications

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Mosconi, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy